CLINICAL TRIAL: NCT04839562
Title: Solriamfetol for ADHD in Adults: A Double-Blind Placebo Controlled Pilot Study
Brief Title: A Controlled Study of Solriamfetol for Attention Deficit Hyperactivity Disorder (ADHD) in Adults
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Craig B. Surman, MD, Scientific Coordinator, Adult ADHD Research Program, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020P003608
Record Dates: First submitted 2021-04-06; First posted 2021-04-09 (Actual); Results first posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: attention deficit hyperactivity disorder; clinical trial; solriamfetol
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — solriamfetol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- solriamfetol (Experimental): Participant will receive daily doses of solriamfetol, at 75 mg at week one and 150 mg at week 2, and with intention that dosing remain stable for the last four weeks of study participation, such that investigators will ask a subject to go back down to 75 mg during any of the weeks following week 2 only if only if 150 mg is not tolerated.
  Interventions: Drug: Solriamfetol 75 MG; Drug: Solriamfetol 150 MG
- placebo (Placebo Comparator): Participant will receive daily doses of placebo, at 75 mg at week one and 150 mg at week 2, and with intention that dosing remain stable for the last four weeks of study participation, such that investigators will ask a subject to go back down to 75 mg during any of the weeks following week 2 only if only if 150 mg is not tolerated.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Solriamfetol 75 MG — Daily oral consumption
  Other Names: Sunosi 75 mg
  Arms: solriamfetol
Drug: Solriamfetol 150 MG — Daily oral consumption
  Other Names: Sunosi 150 mg
  Arms: solriamfetol
Other: Placebo — Placebo
  Arms: placebo

SUMMARY:
A double-blind, placebo controlled study of solriamfetol for adults age 18 to 65 with diagnosis of Attention Deficit Hyperactivity Disorder.

DETAILED DESCRIPTION:
Subjects will be between 18 and 65 years old, have at least 5 current symptoms of inattentive or impulsive-hyperactive traits, and childhood onset of ADHD symptoms, defined as two symptoms of inattentive or of impulsive/hyperactive traits by the age of 12. Subjects will also have a score of 20 or more on the Adult ADHD Investigator Symptom Report Scale (AISRS).

The investigators will exclude individuals who are contraindicated by current FDA label recommendations, which elaborates appropriate use of solriamfetol for individuals with sleep apnea and narcolepsy.

This will be a a six week, double blind, dose-optimization study. After giving informed consent to participate, participants will undergo a comprehensive assessment including a psychiatric assessment reviewing eligibility.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ages 18-65 years of age.
2. A diagnosis of childhood-onset ADHD, meeting the Diagnostic and Statistical Manual-5 (DSM-5) criteria for ADHD in adulthood, including at least 5 current symptoms of inattentive or impulsive-hyperactive traits, and childhood onset by age 12, defined as two symptoms of inattentive or of impulsive/hyperactive traits by the age of 12.
3. A score of 20 or more on the Adult ADHD Investigator Symptom Report Scale (AISRS)

Exclusion Criteria:

1. Individuals with known renal insufficiency or renal impairment.
2. A history of intolerance to solriamfetol
3. Pregnant or nursing females, and individuals unwilling to use adequate contraceptive methods to avoid conception while they are receiving study agent and for 1 month after the last dose of study agent. For female subjects of childbearing potential adequate contraceptive methods will include: a medically acceptable form of birth control (such as male or female condoms with or without spermicidal agent, diaphragm or cervical cap with spermicide, medically prescribed IUD, hormonal contraceptives like birth control pills, or abstinence). For male subjects this will include use of male condom, being status post vasectomy at least 4 months prior to initiation of study drug exposure, or abstinence during the study.
4. A known unstable major medical illness including hepatic, renal, gastroenterological, respiratory, cardiovascular (including hypertension ≥ 140/90 mmHg), endocrinologic (e.g. thyroid), neurologic (e.g. seizure), immunologic, hematologic, or psychiatric (including an active substance use disorder, psychosis, bipolar disorder, major depression) disorder.
5. Any medical condition that the Principal Investigator (PI) believes will be exacerbated by study participation.
6. A history of cancer (except localized skin cancer without metastases or in situ cervical cancer) within 5 years prior to screening.
7. A known history of narrow-angle glaucoma.
8. Current (within 3 months) DSM-V criteria for abuse or dependence with any psychoactive substance other than nicotine.
9. Multiple adverse drug reactions, defined as previous moderate to severe adverse experiences while on two or more chemically unrelated compounds, where these reactions were unpredictable from the known pharmacology of the drug.
10. Any other concomitant medication with primarily central nervous system activity that are catecholaminergic such as stimulants or atomoxetine, or have strong noradrenergic mechanisms of action such as duloxetine or venlafaxine or buproprion. Subjects may be included who are taking stable doses of agents with primary serotonergic (such as selective serotonin reuptake inhibitors or buspirone), gabaergic (such as gabapentin, pregabalin), or other anticonvulsants. We will also allow participation by individuals with rare (predicted to be less than twice a week) use of prn benzodiazepines or sedative-hypnotics.
11. Current use of MAO Inhibitor or use within the past two weeks.
12. Concomitant medications with high potential for dopaminergic or sympathomimetic effects.
13. Investigator and his/her immediate family; defined as the investigator's spouse, parent, child, grandparent, or grandchild.

14, Reasonable suspicion of inability, in the judgement of the investigator, to appropriately monitor experiences during the study and take steps to report these experiences or respond in a manner preserving personal health and safety.

15. If clinically appropriate, any subjects taking medication exclusionary to the study (including agents used for management of ADHD) must be tapered off this medication prior to baseline visit for the length of 5 half-lives of the medication, corresponding to 95% of the agent leaving the participant's system), plus several days or otherwise sufficient period of time to allow assessment of eligibility for participation off medication.

16. Any condition, including a moderate to severe untreated sleep disorder or other mental health disorder, that renders inability, in the investigator's judgement, to determine whether ADHD symptoms are primarily due to ADHD.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-08-06 (Actual); Primary Completion 2023-01-27 (Actual); Study Completion 2023-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Surman, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Surman CBH, Walsh DM, Horick N, DiSalvo M, Vater CH, Kaufman D. Solriamfetol for Attention-Deficit/Hyperactivity Disorder in Adults: A Double-Blind Placebo-Controlled Pilot Study. J Clin Psychiatry. 2023 Oct 9;84(6):23m14934. doi: 10.4088/JCP.23m14934. PMID 37819836

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 66 participants signed consent to participate in the study, per definition of enrollment. 6 of these participants ended up being excluded, and were never exposed (3 lost to follow up, 2 withdrew, 1 found to be ineligible after enrollment). 60 participants total were exposed to solriamfetol or placebo.
Period: Overall Study
Arm/Group | Solriamfetol | Placebo
Started | 29 | 31
Completed | 29 | 29
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Solriamfetol | Placebo | Total
Number analyzed (Participants) | 29 | 31 | 60
Age, Continuous [Mean (Full Range); unit: years] | 36.2 [19 to 61] | 36.9 [22 to 60] | 36.6 [19 to 61]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 10 | 17 | 27
  Female | 17 | 12 | 29
  Other | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 6
  Not Hispanic or Latino | 25 | 29 | 54
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 5 | 2 | 7
  Black or African American | 2 | 2 | 4
  White | 19 | 25 | 44
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Highest Education [Count of Participants; unit: Participants]
  High School Graduate | 1 | 0 | 1
  Some college but no college degree | 4 | 2 | 6
  Associate's Degree | 2 | 3 | 5
  Bachelor's or RN Degree | 10 | 16 | 26
  Some graduate school but no graduate degree | 2 | 2 | 4
  Master's Degree | 3 | 2 | 5
  Doctoral or Law Degree | 7 | 6 | 13
Marital Status [Count of Participants; unit: Participants]
  Married | 13 | 12 | 25
  Unmarried | 16 | 19 | 35
Socioeconomic Status [Mean (Standard Deviation); unit: Dollars] — Yearly Household Income
  Dollars | 98349 (31349) | 119593 (33612) | 109325 (34041)
Clinical Global Impressions Severity (Baseline) [Count of Participants; unit: Participants] — Clinical Global Impressions (CGI) scale for ADHD. The CGI is a measure of illness severity, improvement, and efficacy of treatment. The CGI asks the clinician one question: "Considering your total clinical experience with this particular population, how mentally ill is the patient at this time?" A higher number signifies a higher rating of mental illness.
  Participants
    4 Moderately Ill | 22 | 25 | 47
    5 Markedly Ill | 7 | 6 | 13
Global Assessment of Functioning Scale Score (Baseline) [Mean (Full Range); unit: total score on a scale] — The Global Assessment of Functioning (GAF) scale is a clinician rated scale that assesses global functioning using a scale from 1 (worst) to 100 (best).
  total score on a scale | 63.8 [60 to 68] | 63.8 [61 to 66] | 63.8 [60 to 68]

OUTCOME MEASURES:

1. Primary Outcome: Adult Attention Deficit Hyperactivity Disorder (ADHD) Investigator Symptom Rating Scale (AISRS) Total Score
Description: Difference between active and placebo for change in Adult ADHD Investigator Symptom Rating total score from baseline to week 6 visit. The minimum score on this scale is 0, the maximum score for the scale is 54 points.Higher numbers indicate more ADHD symptoms, lower scores reflect lower ADHD symptoms.
Time Frame: six weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Solriamfetol | Placebo
Number analyzed (Participants) | 29 | 31
score on a scale | -7.6 [-9.9 to -5.3] | -2.1 [-4.4 to 0.2]
Statistical Analysis 1: Comparison: Solriamfetol vs Placebo; Test type: Superiority; p = .0106, t-test, 2 sided; Mean Difference (Final Values) = -4.3, 95% CI 2-sided [-7.7 to -1]

2. Primary Outcome: A Priori Definition of Clinical Improvement
Description: 25% reduction in ADHD symptoms as measured by the Adult ADHD Investigator Symptom Rating Scale (AISRS), and a Clinical Global Impression Improvement score of 2 (much) or 1 (very much) improved. The minimum score on the AISRS scale is 0, the maximum score for the scale is 54 points.Higher numbers indicate more ADHD symptoms, lower scores reflect lower ADHD symptoms. The Clinical Global Impression (CGI) Improvement scores range from 0 to 7, with 0=not assessed,1=very much improved), 2=much improved, through to 7=very much worse. Lower scores therefore mean better outcomes.
Time Frame: six weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Solriamfetol | Placebo
Number analyzed (Participants) | 29 | 31
Participants | 13 | 2
Statistical Analysis 1: Comparison: Solriamfetol vs Placebo; Test type: Superiority; p = .002, Fisher Exact

3. Secondary Outcome: Number of Participants Reaching 0.5 Standard Deviation Improvement on Brief Rating Inventory of Executive Function-Adult Version (BRIEF-A): Global Executive Composite Index
Description: We secondarily will explore whether there are reduced symptoms of executive dysfunction (defined by a 0.5 standard deviation improvement on the Brief Rating Inventory of Executive Function-Adult Version (BRIEF-A) self-report total (GEC). The BRIEF has 75 items that are rated in terms of frequency on a 3-point scale: 0 (never), 1 (sometimes), 2 (often). The range of scores is 0 to 225. Ther are 9 subscales that are indexed under two categories, Behavioral Regulation (BRI) and Metacognition (MI), and these indexes form the overall summary score, the Global Executive Composite (GEC). Raw scores for each scale are summed and T scores (M = 50, SD = 10) are used to interpret the individual's level of executive functioning. Higher scores reflect worse functioning, and lower scores reflect better functioning.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Solriamfetol | Placebo
Number analyzed (Participants) | 29 | 29
Participants | 20 | 10
Statistical Analysis 1: Comparison: Solriamfetol vs Placebo; Test type: Superiority; p = .0173, Fisher Exact

4. Secondary Outcome: Number of Participants Reaching 0.5 Standard Deviation Improvement on Brief Rating Inventory of Executive Function-Adult Version (BRIEF-A): Behavioral Regulation Index
Description: We secondarily will explore whether there are reduced symptoms of executive dysfunction (defined by a 0.5 standard deviation improvement on the Brief Rating Inventory of Executive Function-Adult Version (BRIEF-A) self-report total (GEC) or subscale scores. The BRIEF has 75 items that are rated in terms of frequency on a 3-point scale: 0 (never), 1 (sometimes), 2 (often). The range of scores is 0 to 225. There are 9 subscales that are indexed under two categories, one of which is Behavioral Regulation (BRI). The raw score of the BRI is converted into a T scores (M = 50, SD = 10) are used to interpret the individual's level of executive functioning. Higher scores reflect worse functioning, and lower scores reflect better functioning.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Solriamfetol | Placebo
Number analyzed (Participants) | 29 | 29
Participants | 18 | 11
Statistical Analysis 1: Comparison: Solriamfetol vs Placebo; Test type: Superiority; p = .1144, Fisher Exact

5. Secondary Outcome: Number of Participants Reaching 0.5 Standard Deviation Improvement on Brief Rating Inventory of Executive Function-Adult Version (BRIEF-A): Metacognition Index
Description: We secondarily will explore whether there are reduced symptoms of executive dysfunction (defined by a 0.5 standard deviation improvement on the Brief Rating Inventory of Executive Function-Adult Version (BRIEF-A) self-report total (GEC) or subscale scores). The BRIEF has 75 items that are rated in terms of frequency on a 3-point scale: 0 (never), 1 (sometimes), 2 (often). The range of scores is 0 to 225. There are 9 subscales that are indexed under two categories, one of which is Metacognition Index (MI). The raw score of the MI is converted into a T scores (M = 50, SD = 10) are used to interpret the individual's level of executive functioning. Higher scores reflect worse functioning, and lower scores reflect better functioning.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Solriamfetol | Placebo
Number analyzed (Participants) | 29 | 29
Participants | 19 | 10
Statistical Analysis 1: Comparison: Solriamfetol vs Placebo; Test type: Superiority; p = .0348, Fisher Exact

6. Secondary Outcome: Number of Participants Reaching 0.5 Standard Deviation Improvement on Brief Rating Inventory of Executive Function-Adult Version (BRIEF-A): Inhibit Subscale
Description: We secondarily will explore whether there are reduced symptoms of executive dysfunction (defined by a 0.5 standard deviation improvement on the Brief Rating Inventory of Executive Function-Adult Version (BRIEF-A) self-report total (GEC) or subscale scores). The BRIEF has 75 items that are rated in terms of frequency on a 3-point scale: 0 (never), 1 (sometimes), 2 (often). The range of scores is 0 to 225. There are 9 subscales, one of which is the Inhibit subscale. Raw scores for this scale are summed and T scores (M = 50, SD = 10) are used to interpret the individual's level of executive functioning. Higher scores reflect worse functioning, and lower scores reflect better functioning.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Solriamfetol | Placebo
Number analyzed (Participants) | 29 | 29
Participants | 11 | 10
Statistical Analysis 1: Comparison: Solriamfetol vs Placebo; Test type: Superiority; p = 1, Fisher Exact

7. Secondary Outcome: Number of Participants Reaching 0.5 Standard Deviation Improvement on Brief Rating Inventory of Executive Function-Adult Version (BRIEF-A): Shift Subscale
Description: We secondarily will explore whether there are reduced symptoms of executive dysfunction (defined by a 0.5 standard deviation improvement on the Brief Rating Inventory of Executive Function-Adult Version (BRIEF-A) self-report total (GEC) or subscale scores). The BRIEF has 75 items that are rated in terms of frequency on a 3-point scale: 0 (never), 1 (sometimes), 2 (often). The range of scores is 0 to 225. Ther are 9 subscales that are indexed under two categories, one of which is the Shift subscale. Raw scores for this scale are summed and T scores (M = 50, SD = 10) are used to interpret the individual's level of executive functioning. Higher scores reflect worse functioning, and lower scores reflect better functioning.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Solriamfetol | Placebo
Number analyzed (Participants) | 29 | 29
Participants | 20 | 10
Statistical Analysis 1: Comparison: Solriamfetol vs Placebo; Test type: Superiority; p = .0173, Fisher Exact

8. Secondary Outcome: Number of Participants Reaching 0.5 Standard Deviation Improvement on Brief Rating Inventory of Executive Function-Adult Version (BRIEF-A): Emotional Control Subscale
Description: We secondarily will explore whether there are reduced symptoms of executive dysfunction (defined by a 0.5 standard deviation improvement on the Brief Rating Inventory of Executive Function-Adult Version (BRIEF-A) self-report total (GEC) or subscale scores). The BRIEF has 75 items that are rated in terms of frequency on a 3-point scale: 0 (never), 1 (sometimes), 2 (often). The range of scores is 0 to 225. There are 9 subscales, one of which is the Emotional Control subscale. Raw scores for this scale are summed and T scores (M = 50, SD = 10) are used to interpret the individual's level of executive functioning. Higher scores reflect worse functioning, and lower scores reflect better functioning.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Solriamfetol | Placebo
Number analyzed (Participants) | 29 | 29
Participants | 16 | 10
Statistical Analysis 1: Comparison: Solriamfetol vs Placebo; Test type: Superiority; p = .1864, Fisher Exact

9. Secondary Outcome: Number of Participants Reaching 0.5 Standard Deviation Improvement on Brief Rating Inventory of Executive Function-Adult Version (BRIEF-A): Self-Monitor Subscale
Description: We secondarily will explore whether there are reduced symptoms of executive dysfunction (defined by a 0.5 standard deviation improvement on the Brief Rating Inventory of Executive Function-Adult Version (BRIEF-A) self-report total (GEC) or subscale scores). The BRIEF has 75 items that are rated in terms of frequency on a 3-point scale: 0 (never), 1 (sometimes), 2 (often). The range of scores is 0 to 225. There are 9 subscales, one of which is the Self-Monitor subscale. Raw scores for this scale are summed and T scores (M = 50, SD = 10) are used to interpret the individual's level of executive functioning. Higher scores reflect worse functioning, and lower scores reflect better functioning.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Solriamfetol | Placebo
Number analyzed (Participants) | 29 | 29
Participants | 13 | 9
Statistical Analysis 1: Comparison: Solriamfetol vs Placebo; Test type: Superiority; p = .4173, Fisher Exact

10. Secondary Outcome: Number of Participants Reaching 0.5 Standard Deviation Improvement on Brief Rating Inventory of Executive Function-Adult Version (BRIEF-A): Initiate Subscale
Description: We secondarily will explore whether there are reduced symptoms of executive dysfunction (defined by a 0.5 standard deviation improvement on the Brief Rating Inventory of Executive Function-Adult Version (BRIEF-A) self-report total (GEC) or subscale scores). The BRIEF has 75 items that are rated in terms of frequency on a 3-point scale: 0 (never), 1 (sometimes), 2 (often). The range of scores is 0 to 225. There are 9 subscales, one of which is the Initiate subscale. Raw scores for this scale are summed and T scores (M = 50, SD = 10) are used to interpret the individual's level of executive functioning. Higher scores reflect worse functioning, and lower scores reflect better functioning.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Solriamfetol | Placebo
Number analyzed (Participants) | 29 | 29
Participants | 18 | 9
Statistical Analysis 1: Comparison: Solriamfetol vs Placebo; Test type: Superiority; p = .0343, Fisher Exact

11. Secondary Outcome: Number of Participants Reaching 0.5 Standard Deviation Improvement on Brief Rating Inventory of Executive Function-Adult Version (BRIEF-A): Working Memory Subscale
Description: We secondarily will explore whether there are reduced symptoms of executive dysfunction (defined by a 0.5 standard deviation improvement on the Brief Rating Inventory of Executive Function-Adult Version (BRIEF-A) self-report total (GEC) or subscale scores) The BRIEF has 75 items that are rated in terms of frequency on a 3-point scale: 0 (never), 1 (sometimes), 2 (often). The range of scores is 0 to 225. There are 9 subscales, one of which is the Working Memory subscale. Raw scores for this scale are summed and T scores (M = 50, SD = 10) are used to interpret the individual's level of executive functioning. Higher scores reflect worse functioning, and lower scores reflect better functioning.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Solriamfetol | Placebo
Number analyzed (Participants) | 29 | 29
Participants | 17 | 9
Statistical Analysis 1: Comparison: Solriamfetol vs Placebo; Test type: Superiority; p = .0636, Fisher Exact

12. Secondary Outcome: Number of Participants Reaching 0.5 Standard Deviation Improvement on Brief Rating Inventory of Executive Function-Adult Version (BRIEF-A): Plan/Organize Subscale
Description: We secondarily will explore whether there are reduced symptoms of executive dysfunction (defined by a 0.5 standard deviation improvement on the Brief Rating Inventory of Executive Function-Adult Version (BRIEF-A) self-report total (GEC) or subscale scores). The BRIEF has 75 items that are rated in terms of frequency on a 3-point scale: 0 (never), 1 (sometimes), 2 (often). The range of scores is 0 to 225. There are 9 subscales, one of which is the Plan/Organize subscale. Raw scores for this scale are summed and T scores (M = 50, SD = 10) are used to interpret the individual's level of executive functioning. Higher scores reflect worse functioning, and lower scores reflect better functioning.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Solriamfetol | Placebo
Number analyzed (Participants) | 29 | 29
Participants | 19 | 11
Statistical Analysis 1: Comparison: Solriamfetol vs Placebo; Test type: Superiority; p = .065, Fisher Exact

13. Secondary Outcome: Number of Participants Reaching 0.5 Standard Deviation Improvement on Brief Rating Inventory of Executive Function-Adult Version (BRIEF-A): Task Monitor Subscale
Description: We secondarily will explore whether there are reduced symptoms of executive dysfunction (defined by a 0.5 standard deviation improvement on the Brief Rating Inventory of Executive Function-Adult Version (BRIEF-A) self-report total (GEC) or subscale scores). The BRIEF has 75 items that are rated in terms of frequency on a 3-point scale: 0 (never), 1 (sometimes), 2 (often). The range of scores is 0 to 225. There are 9 subscales, one of which is the Task Monitor subscale. Raw scores for this scale are summed and T scores (M = 50, SD = 10) are used to interpret the individual's level of executive functioning. Higher scores reflect worse functioning, and lower scores reflect better functioning.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Solriamfetol | Placebo
Number analyzed (Participants) | 29 | 29
Participants | 18 | 11
Statistical Analysis 1: Comparison: Solriamfetol vs Placebo; Test type: Superiority; p = .1144, Fisher Exact

14. Secondary Outcome: Number of Participants Reaching 0.5 Standard Deviation Improvement on Brief Rating Inventory of Executive Function-Adult Version (BRIEF-A): Organization of Materials Subscale
Description: We secondarily will explore whether there are reduced symptoms of executive dysfunction (defined by a 0.5 standard deviation improvement on the Brief Rating Inventory of Executive Function-Adult Version (BRIEF-A) self-report total (GEC) or subscale scores). The BRIEF has 75 items that are rated in terms of frequency on a 3-point scale: 0 (never), 1 (sometimes), 2 (often). The range of scores is 0 to 225. There are 9 subscales, one of which is the Organization of Materials subscale. Raw scores for this scale are summed and T scores (M = 50, SD = 10) are used to interpret the individual's level of executive functioning. Higher scores reflect worse functioning, and lower scores reflect better functioning.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Solriamfetol | Placebo
Number analyzed (Participants) | 29 | 29
Participants | 14 | 9
Statistical Analysis 1: Comparison: Solriamfetol vs Placebo; Test type: Superiority; p = .2829, Fisher Exact

ADVERSE EVENTS:
Time Frame: Baseline to endpoint (6 weeks)
Description: Adverse events were reported at weekly study visits or spontaneously by subjects
Arm/Group | Solriamfetol | Placebo
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/31
Other Adverse Events (participants affected / at risk) | 28/29 | 28/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Solriamfetol (N=29) | Placebo (N=31)
Cold/Infection/Allergy (Infections and infestations) | 13 | 17
Increased Appetite (Metabolism and nutrition disorders) | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 5 | 2
Headache (General disorders) | 14 | 9
Nausea/Vomiting/Diarrhea (Gastrointestinal) (Gastrointestinal disorders) | 7 | 2
Insomnia (General disorders) | 9 | 5
Sedation (General disorders) | 3 | 1
Increased Energy (General disorders) | 4 | 1
Cardiovascular (Cardiac disorders) | 5 | 1
Tense/jittery (General disorders) | 1 | 0
Agitated/irritable (General disorders) | 3 | 2
Anxious/Worried (Psychiatric disorders) | 0 | 1
Mucosal Dryness (Gastrointestinal disorders) | 3 | 4
Dizzy/Lightheaded (General disorders) | 1 | 0
Neurological (Nervous system disorders) | 4 | 1
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 7 | 7
Genitourinary (Renal and urinary disorders) | 3 | 2
Dermtological (Skin and subcutaneous tissue disorders) | 1 | 4
Other (General disorders) | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-22): https://cdn.clinicaltrials.gov/large-docs/62/NCT04839562/Prot_SAP_000.pdf